CLINICAL TRIAL: NCT03644316
Title: BandGrip® Closure of Surgical Incisions Following Arthroscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BandGrip (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPS-002
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BandGrip (Experimental): Topical skin closure device
  Interventions: Device: BandGrip skin closure device

INTERVENTIONS:
Device: BandGrip skin closure device — topical skin closure device

SUMMARY:
A single-arm, prospective, unblinded, post marketing, single center study using BandGrip to close incisions post arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
The study objective is to assess the ease of incision closure, the cosmetic appearance of the wounds on follow-up, and general subject satisfaction with the appearance of the healed incisions following use of BandGrip. Up to 25 subjects will be enrolled at a single center.

Subjects who have undergone arthroscopic surgery of the shoulder and require closure of one or two skin puncture sites will be enrolled. Following incision closure subjects will be seen at the time of BandGrip removal (approximately 7-14 days after closure) and at 30 days for assessment of the incisions.

The incidence of wound closure for each treated puncture site, defined as continuous approximation of wound margins from the time of wound closure until the day of removal of the wound closure device without dehiscence or need for reclosure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is ≥ 18 years of age. 2. Subject had an arthroscopic shoulder procedure and has at least two skin incisions that are assessed as requiring temporary approximation of the skin edges.

  3. The length of the subject's surgical incisions is less than or equal to 1.5 inches.

  4. Subject must be willing to follow instructions for wound care provided by investigator and refrain from picking at the treatment device, applying topical medications to the wound, and swimming or soaking in a tub until the wound closure device is removed.

  5. Subject agrees to return for all required follow-up evaluations. 6. Subject is able to comprehend and give informed consent for participation in this study.

Exclusion Criteria:

* 1. Subject has a recent history of bleeding, coagulation, and/or clotting disorders.

  2. Subject is on dialysis. 3. Subject has a history of inflammatory and/or allergic diseases or conditions of the skin involving the location of the incisions (e.g., psoriasis, Eczema, or dermatitis).

  4. Subject has a history of drug abuse. 5. Subject has a history of chronic use of oral steroids or immunosuppressants. 6. Subject has known personal or family history of keloid or hypertrophic scarring.

  7. Subject has a history of abnormal wound healing. 8. Subject's incisions are in a high skin tension area. 9. Subject has a known allergy to BandGrip material (polycarbonate). 10. Subject has a known cognitive or psychiatric disorder. 11. Subject has an incision at site of active rash/skin lesion making evaluation difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of complete would closure | 30 days post treatment
  complete approximation of wound margins from the time of wound closure until the day of removal of the wound closure device without dehiscence or need for reclosure.

SECONDARY OUTCOMES:
Incidence of partial wound apposition | 10 and 30 days post closure
  at least 50% wound apposition
Incision Cosmesis | 10 and 30 days post closure
  use of a 0 to 100 mm visual analog scale (100mm is best outcome)
Subject Satisfaction with cosmetic appearance of healed incision | 10 and 30 days post surgery
  use of a 0 to 100mm visual analog scale (100mm is best outcome)
Physician Satisfaction with cosmetic appearance of healed incision | 10 and 30 days post surgery
  use of a 0 to 100mm visual analog scale (100mm is best outcome)
Time to closure and removal of wound closure device | at surgical procedure and 10 days
  amount of time to apply and remove BandGrip
Adverse events | 30 days post surgery
  collection of device complaints

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Galles, MD, Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No